CLINICAL TRIAL: NCT05964166
Title: Tetragraph® Monitor: Tolerance of Preoperative Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chief of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003295
Record Dates: First submitted 2023-06-02; First posted 2023-07-27 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Tetragraph (Experimental)
  Interventions: Device: TetraGraph NMT Monitor

INTERVENTIONS:
Device: TetraGraph NMT Monitor — TetraGraph is a unique, EMG=based portable device for quantitative (objective) monitoring of neuromuscular function. It is a precise and easy to use tool for monitoring depth of block, ensuring adequate recovery of muscle function, and aiding the clinician to reduce the incidence of residual block.

SUMMARY:
This is a prospective, non-blinded, single arm study. The primary objective of this study is to evaluate the tolerance to preoperative placement of the adhesive sensor for the Tetragraph® Neuromuscular Transmission Monitor in pediatric-sized patients ≤ 12 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring anesthetic care and use of neuromuscular blockade
2. Age ≤ 12 years
3. ASA 1-4

Exclusion Criteria:

1. History of a peripheral neurologic or neuropathic disorder
2. Upper extremity cannot be used for TOF monitoring
3. Undergoing a surgical procedure in which neuromuscular blockade is not required
4. Patient is edematous
5. Patients with significant behavioral or neurocognitive issues which affect behavior and impact the ability to place the sensor

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulled Off Sensor: Patients that pulled off the TetraGraph sensor before arrival to the OR.
- Sensor Intact: Patients that arrived to the OR with the sensor intact and functioning.
Period: Overall Study
Arm/Group | Pulled Off Sensor | Sensor Intact
Started | 14 | 26
Completed | 14 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulled Off Sensor | Sensor Intact | Total
Number analyzed (Participants) | 14 | 26 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 26 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 0.98 [0.61 to 4.89] | 5.24 [0.77 to 8.71] | 3.70 [0.72 to 7.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 11 | 20 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 25 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 11 | 19 | 30
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 26 | 40
Weight (kg) [Median (Inter-Quartile Range); unit: kilograms] | 9.88 [7.35 to 16.9] | 20 [8.99 to 27.4] | 15.55 [8.27 to 25.35]
Height (cm) [Median (Inter-Quartile Range); unit: centimeters] | 73.5 [62 to 111.9] | 110.2 [74 to 130.3] | 103 [70 to 125.5]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 17.81 [16.33 to 19] | 15.8 [14.71 to 18.15] | 16.4 [15.16 to 18.58]
ASA physical status [Count of Participants; unit: Participants] — American Society of Anesthesiologists classification system is to assess and communicate a patient's pre-anesthesia medical co-morbidities. ASA 1 = healthy patient, 2 = mild systemic disease, 3 = severe systemic disease, 4 = severe systemic disease that is a constant threat to life.
  Participants
    ASA I | 3 | 11 | 14
    ASA II | 8 | 10 | 18
    ASA III | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Tolerance to Preop Placement as Assessed by Likert Scale
Description: Patient's tolerance to preoperative placement of the adhesive sensor for the Tetragraph® Neuromuscular Transmission Monitor will be assessed by using a 10-point Likert scale with 0=very badly/pulled sensor off and 10=very well/left sensor alone.
Time Frame: 30 mins. prior to surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale (0-10)
Arm/Group | Pulled Off Sensor | Sensor Intact
Number analyzed (Participants) | 14 | 26
units on a scale (0-10)
  Research team member assessment | 0 [0 to 0] | 10 [9 to 10]
  Family member assessment | 0 [0 to 0] | 10 [10 to 10]

2. Secondary Outcome: Application Ease
Description: The ease of preoperative placement of the adhesive sensor for the Tetragraph® Neuromuscular Transmission Monitor will be assessed by the research staff by using a 10-point Likert scale with 0=very difficult and 10=very easy.
Time Frame: 30 minutes prior to surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale (0-10)
Arm/Group | Pulled Off Sensor | Sensor Intact
Number analyzed (Participants) | 14 | 26
units on a scale (0-10) | 4 [0 to 10] | 10 [7 to 10]

ADVERSE EVENTS:
Time Frame: Day of surgery
Arm/Group | Pulled Off Sensor | Sensor Intact
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/26
Other Adverse Events (participants affected / at risk) | 0/14 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT05964166/Prot_001.pdf
  • Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT05964166/SAP_002.pdf